CLINICAL TRIAL: NCT02178072
Title: A Window Study to Assess the Activity of Demethylation Therapy in Patients With HPV-Positive Compared With HPV-Negative Head and Neck Squamous Cell Carcinoma, With Response Assessment and Biomarker Expansion Cohort in HPV-Positive Oropharynx Cancer
Brief Title: Window Trial 5-aza in HNSCC, T-tare
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404013771
Record Dates: First submitted 2014-06-23; First posted 2014-06-30 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPV positive (Other): HPV positive patients
  Interventions: Drug: 5-Azacitadine
- HPV negative (Other): HPV negative patients
  Interventions: Drug: 5-Azacitadine

INTERVENTIONS:
Drug: 5-Azacitadine
  Other Names: Vidaza

SUMMARY:
The purpose of this study is to assess the activity of 5-azacitidine in patients with Human Papilloma Virus (HPV)-positive and HPV- negative head and neck squamous cell carcinoma (HNSCC). The response activity will be determined by analyzing your tumor tissue prior to and after treatment with 5-azacitidine. Preliminary studies in mice bearing human head and neck cancers or head and neck cancer cells cultured in laboratories suggest that treatment with 5-azacitidine increases changes in cancer cells that lead to their death. This study is designed to determine if similar changes occur in cancer cells of patients with head and neck cancer.

The study also aims to determine the amount of a specific type of protein, p53 before and after treatment. Research has shown that the p53 protein is associated with anti-tumor activity.

Finally, this study is measuring the amount of a specific type of protein called interferon in your tumor tissue. Interferons are proteins made and released by the body in response to pathogens (disease causing agents) such as viruses, bacteria, or tumor cells. Interferons allow for communication between cells to trigger the protective defenses of the immune system that remove pathogens (disease causing agents) or tumors.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objectives of this study are:

• to determine the proportion of HPV-positive patients in whom 5-azacytidine increases APOBEC RNA expression.

Secondary Objectives

The secondary objectives of this study are:

* to investigate response (proliferation, apoptosis), as well as reactivation of IFN pathways in patients treated with 5-azacitadine for HPV-positive and HPV-negative HNSCC.
* to investigate the clinical activity of 5-azacitadine in patients with HPV-positive and HPV-negative HNSCC.
* to investigate the safety of 5-azacitadine in patients with HPV-positive and HPV-negative HNSCC

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed p16 or HPV PCR positive HNSCC with surgically resectable disease
2. Age ≥18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1 or 2
4. ANC greater than or equal to 1500, Hb greater than or equal to 8, platelet count greater than or equal to 100,000

Exclusion Criteria:

1. AST or ALT greater than 2.5 x ULN
2. Known brain metastases
3. Women must not be pregnant or breastfeeding
4. Known allergy to 5-azacitadine
5. Patients receiving any other investigational agents within 4 weeks of starting the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
tumor response | 6 months
  The post-treatment biopsy will occur the day after the last injection of 5-azacytidine. 5-aza is currently FDA-approved and used for therapy of myelodysplastic syndrome. Pre- and post- 5-aza treatment tissue will be analyzed for proliferation (IHC-Ki-67), apoptosis (IHC-cleaved caspase-3, cleaved PARP-1), and for p53 protein (IHC, immunoblots), as well as p53, CDKN1A, MDM2, IFITs, and CCL5 mRNA levels (as described above). The primary outcome is the change from baseline of the p53 protein level in post-treatment vs. pre-treatment biopsies. Although tumor response may not be expected due to the short treatment course, the post-treatment vs. pre-treatment change from baseline of the gross tumor measurements will be used to measure tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burtness, MD, Principal Investigator — Yale University School of Medicine, Smilow Cancer Center at Yale New Haven Hospital, Yale Comprehensive Cancer Center
Locations (1):
- Smilow Cancer Center at Yale New Haven Hospital, New Haven, Connecticut, United States